CLINICAL TRIAL: NCT02349724
Title: A Clinical Research of Chimeric Antigen Receptor(CAR) T Cells Targeting CEA Positive Cancer
Brief Title: A Clinical Research of CAR T Cells Targeting CEA Positive Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Zhi Yang, Researcher of Biotherpy Center, Southwest Hospital, China
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMMU-BTC-002
Record Dates: First submitted 2015-01-25; First posted 2015-01-29 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2016-03

CONDITIONS: Lung Cancer; Colorectal Cancer; Gastric Cancer; Breast Cancer; Pancreatic Cancer
Keywords: CEA; CAR T
MeSH Terms: conditions — Lung Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Breast Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Pancreatic cancer (Other): Pancreatic cancer treated with Anti-CEA-CAR T.
  Interventions: Biological: Anti-CEA-CAR T
- Lung cancer (Other): Lung cancer treated with T cells modified with Anti-CEA-CAR T.
  Interventions: Biological: Anti-CEA-CAR T
- Gastric cancer (Other): Gastric cancer treated with T cells modified with Anti-CEA-CAR T.
  Interventions: Biological: Anti-CEA-CAR T
- Breast cancer (Other): Breast cancer treated with T cells modified with Anti-CEA-CAR T.
  Interventions: Biological: Anti-CEA-CAR T
- Colorectal cancer (Other): Colorectal cancer treated with T cells modified with Anti-CEA-CAR T.
  Interventions: Biological: Anti-CEA-CAR T

INTERVENTIONS:
Biological: Anti-CEA-CAR T — T cells modified with CEA targeted chimeric antigen receptor.

SUMMARY:
The main purpose of this research is to verify the safety of CEA targeted chimeric antigen receptor T cells and to determine the proper dosage of CAR T cells infused.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR)-modified T cells have demonstrated great successes in treating even late stage cluster of differentiation antigen 19 (CD19) positive B cell malignancies. But it has not yet been fully explored in solid tumors. The carcino-embryonic antigen(CEA) is widely expressed in cancers like gastric cancer, lung cancer, pancreatic cancer, breast cancer and colorectal cancer. To confirm if CAR T cells still function in solid tumors, we have developed anti-CEA CAR-modified T cells. Preclinical studies have demonstrated effective killing of CEA target cells. In this study, the CEA CARs, will be evaluated in CEA positive gastric cancer, lung cancer, pancreatic cancer, breast cancer and colorectal cancer patients. The primary goal is to confirm its adverse effects including cytokine storm response and any other adverse effects. In addition, tumor targeting and disease status after treatment will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory CEA positive lung cancer, pancreatic cancer, gastric cancer, breast cancer and colorectal cancer.
2. KPS>60.
3. Life expectancy>3 months.
4. Gender unlimited, age from 18 years to 80 years.
5. Disease progresses but reserves reaction to recent treatments.
6. Patients who have failed at least one line of a standard treatment.
7. No serious mental disorder.
8. Patients must have adequate cardiac function(no cardiac disease, LVEF≥40% ), adequate pulmonary function as indicated by room air oxygen saturation of >94%, and adequate renal function(Cr≤133umol/L).
9. No other serious diseases(autoimmune disease, immunodeficiency etc.).
10. No other tumors.
11. Patients volunteer to participate in the research.

Exclusion Criteria:

1. KPS<50.
2. Patients are allergic to cytokines.
3. MODS.
4. Uncontrolled active infection.
5. Acute or chronic GVHD.
6. Treated with T cell inhibitor.
7. Pregnancy and nursing females.
8. HIV affected.
9. Other situations we think improper for the research.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2014-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events of each patient. | 3 years
  Determine the toxicity profile of the CEA targeted CAR T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Survival time of Anti-CEA CAR T cells in vivo. | 3 years
  To evaluate the presence of circulating CAR T cells with flow cytometry and real time PCR in patient blood.
Efficacy of anti-CEA CAR T cells to confirm the ability of CAR T cells to kill CEA positive cancer cells | 12 weeks
Maximum tolerated dose (MTD) of CEA targeted CAR T cells. | 4 weeks
  To confirm the maximum tolerated dose of CEA targeted CAR T cells.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Qian, MD, PhD, Study Chair — Southwest Hospital, China
Locations (1):
- Southwest Hospital of Third Millitary Medical University, Chongqing, Chongqing Municipality, China